CLINICAL TRIAL: NCT02444936
Title: A Pilot Study Using a Randomized Design to Evaluate the Immunologic Efficacy and Safety of ZOSTAVAX in Persons Imminently Receiving Chemotherapy for Solid Organ Tumors
Brief Title: ZOSTAVAX in Persons Imminently Receiving Chemotherapy for Solid Organ Tumors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, David Canaday, Associate Director of Research, GRECC, Louis Stokes VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Canaday Zostavax
Record Dates: First submitted 2015-05-07; First posted 2015-05-15 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Shingles
Keywords: solid tumor; chemotherapy; vaccine
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZOSTAVAX (Active Comparator): ZOSTAVAX shingles vaccine Zoster vaccine live Single 0.65mL subcutaneous injection
  Interventions: Drug: ZOSTAVAX
- Control (No Intervention): There is no drug given in this arm.

INTERVENTIONS:
Drug: ZOSTAVAX — Shingles vaccine
  Other Names: Voster vaccine live
  Arms: ZOSTAVAX

SUMMARY:
This study evaluates if the shingles vaccine works in those persons that receive it before they receive chemotherapy for solid organ tumors. Half of the participants will receive the ZOSTAVAX shingle vaccine and half of the participants will not received anything.

DETAILED DESCRIPTION:
This study is a single blind randomized clinical trial measuring the immunologic efficacy of ZOSTAVAX vs. no vaccine in 60 adults with solid organ tumors before, during and after chemotherapy. The personnel performing the laboratory studies will be blinded to vaccine vs. no vaccine. In a pilot study of an FDA approved vaccine that is being used within the parameters of the package insert and ACIP recommendations, placebo vaccine is not required to access our key primary immunologic endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ tumor patients that have at least 14 days between entry into the study with ZOSTAVAX vaccination and initial therapy for their malignancy that will include chemotherapy alone or surgery with subsequent chemotherapy plus or minus radiation therapy
* A plan for chemotherapy that at the onset at least an anticipated stop date within 3-6 months of our sample collection phase of the study

Exclusion Criteria:

* Prior history of HZ or shingles vaccine
* Systemic chemotherapy < 3 months prior to enrollment
* Any history of hematologic malignancy, HIV/AIDS, hematopoietic stem cell transplant, or other cellular immunodeficiency state
* Those receiving immunomodulating drugs at the time of vaccination such as prednisone methotrexate, azathioprine, mercaptopurine, or other biologics including TNF-alpha inhibitors
* Widespread metastatic tumor with bone marrow involvement
* Indefinite duration palliative chemotherapy subjects

  * Inability to communicate with the study staff or bring unable to consent for themselves
  * History of anaphylactic/anaphylactiod reaction to gelatin, neomycin, or other components of the vaccine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Canaday, MD, Principal Investigator — Cleveland VA

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ZOSTAVAX | Control
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX | Control | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (6.6) | 64 (9.8) | 64.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Measuring the Efficacy of ZOSTAVAX in Chemotherapy Patients (Changes in ZOSTAVAX-specific IFN-gamma Spot Forming Units Will be Measured by ELISPOT)
Description: To examine the cellular immunologic efficacy as measured by IFN-gamma assays of ZOSTAVAX given to individuals with solid organ tumors at least 14 days prior to initiation of chemotherapy or surgery and then chemotherapy. Changes in ZOSTAVAX-specific IFN-gamma spot forming units will be measured by ELISPOT.
Time Frame: 3 years
Reporting Status: Not Posted

2. Primary Outcome: Measuring the Safety of ZOSTAVAX Given to Chemotherapy Patients (Vaccine Report Card (VRC) to Document Injection-site Adverse Experiences, Systemic Clinical Adverse Experiences (AEs), Concomitant Medications, and Oral Temperatures
Description: To asses the safety of ZOSTAVAX given to subjects that will receive chemotherapy or surgery and then chemotherapy for solid organ tumor at least 14 days after vaccination. Safety and tolerability data will be collected for all subjects throughout the study. Each subject will be given a Vaccine Report Card (VRC) to document injection-site adverse experiences, systemic clinical adverse experiences (AEs), concomitant medications, and oral temperatures (only if feeling feverish) noted during the 14-day post-vaccination period. Participants will be asked to notify the study personnel immediately if any unexpected or serious adverse experience (SAE) occurs. At all study visits subjects will be asked about any unreported SAEs. All AEs and SAEs will be recorded on an AE/SAE case report form and relationship to study vaccine will be determined by the site investigator.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | ZOSTAVAX | Control
Number analyzed (Participants) | 10 | 12
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: We collected the data for the one month after giving the vaccine.
Description: We have the subjects complete a vaccine side effect report card.
Arm/Group | ZOSTAVAX | Control
All-Cause Mortality (participants affected / at risk) | 2/10 | 4/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 2/10 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZOSTAVAX (N=10) | Control (N=12)
mild injection soreness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — mild injection site soreness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2014-10-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT02444936/SAP_000.pdf
  • Informed Consent Form (2014-10-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT02444936/ICF_001.pdf
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT02444936/Prot_002.pdf